CLINICAL TRIAL: NCT02415985
Title: A Pilot Study of the Pharmacokinetics and Safety of Rifabutin 150 mg Once Daily Versus Rifabutin 300 mg Thrice Weekly With Lopinavir/Ritonavir Based HAART in HIV/TB Co-infected Patients
Brief Title: Pharmacokinetics and Safety of Rifabutin 150 mg Once Daily Versus Rifabutin 300 mg Thrice Weekly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Bamrasnaradura Infectious Diseases Institute (Other Government); Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HIV-NAT 116
Record Dates: First submitted 2015-04-01; First posted 2015-04-14 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: HIV; Tuberculosis
Keywords: pharmacokinetics of rifabutin; HIV/TB co-infection; resource limited setting; AUC; Cmax; Cmin; Ctrough
MeSH Terms: conditions — Tuberculosis | interventions — Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rifabutin 150 (Other): rifabutin 150 mg (1 capsule) once daily
  Interventions: Drug: Lopinavir/r will be supplied by NHSO/GPO; Drug: Rifabutin
- rifabutin 300 (Other): rifabutin 150 mg (2 capsules) 300 mg 3 times a week
  Interventions: Drug: Lopinavir/r will be supplied by NHSO/GPO; Drug: Rifabutin

INTERVENTIONS:
Drug: Lopinavir/r will be supplied by NHSO/GPO — 200/50 mg tablet LPV/rtv
  Other Names: LPV/rtv
Drug: Rifabutin

SUMMARY:
To describe the pharmacokinetics of rifabutin 150 mg once daily versus rifabutin 300 mg thrice weekly in combination with LPV/r 400/100mg based HAART in HIV/TB infected patients

DETAILED DESCRIPTION:
The overall aim of the project is to evaluate rifabutin as a replacement for rifampicin, for the combined treatment of tuberculosis and HIV infection. Rifabutin represents an alternative to rifampicin for HIV infected patients as its half-life is longer and the enzymatic induction effect appears to be less important on the associated ART drugs. This phase II trial is to determine precisely the pharmacokinetics parameters of rifabutin in combination with LPV/r regimens in Thai HIV/TB infected patients, in order to define optimal doses that will be further tested in a larger phase III trial comparing safety, tolerability and efficacy of rifabutin and rifampicin regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV positive after voluntary counseling and testing
2. Aged >18-60years of age
3. PI-naïve (NNRTI intolerance/failure) or PI experience ( TB developed during on salvage regimen) without prior PI mutation
4. Any CD4 cell count
5. ALT <5 times ULN
6. Serum creatinine <1.4 mg/dl
7. Hemaglobin >7 mg/L
8. TB is diagnosed and planned to receive stable doses of rifabutin containing anti-TB therapy for at least another 4 week period after initiation of ART
9. No other active OI (CDC class C event), except oral candidiasis or disseminated MAC
10. Body weight >40kg
11. Able to provide written informed consent

Exclusion Criteria:

1. Current use of steroid (except short course steroid for IRIS) and other immunosuppressive agents.
2. Current use of any prohibited medications related to drug pharmacokinetics.
3. Patients with current alcohol or illicit substance use that in the opinion of the site Principal Investigator would conflict with any aspect of the conduct of the trial.
4. Unlikely to be able to remain in follow-up for the protocol defined period.
5. Patients with proven or suspected acute hepatitis. Patients with chronic viral hepatitis are eligible provided ALT, AST < 5 x ULN.
6. Karnofsky performance score <30%
7. TB meningitis and bone/joints ( due to longer period of anti TB drug)
8. Pregnancy
9. Patient choose to use efavirenz, not LPV/r. However, in ART naïve, EFV is allowed after intensive PK of LPV/r and rifabutin at week 2-4.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of rifabutin Cmax | 48 weeks
  Cmax The peak plasma concentration of rifabutin after administration

SECONDARY OUTCOMES:
adverse events | 48 weeks
  number of participants with adverse events
viral load | 48 weeks
CD4 | 48 weeks
  mean CD4 rise from baseline
Monodrug resistant TB | 48 weeks
death | 48 weeks
AIDS event | 48 weeks
TB cure | 48 weeks
TB relapse | 48 weeks
Multidrug-resistant TB (MDR TB) | 48 weeks
TB treatment failure | 48 weeks
Extensively drug resistant TB (XDR TB) | 48 weeks
weight gain | 48 weeks
  change from baseline in weight gain at 48 weeks
defervescence | 48 weeks
  change from baseline in defervescence at 48 weeks
Karnofsky score | 48 weeks
  change from baseline in Karnofsky score at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre
Locations (4):
- Thailand (4):
  - Chest Division, Faculty of Medicine, Chulalongkorn University, Bangkok
  - HIV-NAT, Thai Red Cross - AIDS Research Centre, Bangkok
  - Infectious Diseases, Faculty of Medicine, Chulalongkorn University, Bangkok
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration — http://www.hivnat.org